CLINICAL TRIAL: NCT05995340
Title: An International, Multicenter, Double-blind, Randomized, Parallel-group, Controlled Study to Evaluate the Safety and Effectiveness of ELAPR002f Injectable Gel in Adult Participants With Atrophic Acne Scars
Brief Title: ELAPR002f Injectable Gel in the Treatment of Atrophic Acne Scars
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015-702-008; CIV-23-03-042622 (Other: EUDAMED)
Record Dates: First submitted 2023-08-10; First posted 2023-08-16 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Atrophic Acne Scars
Keywords: Atrophic Acne Scars; ELAPR002f injectable gel

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- ELAPR002f Injectable Gel (Experimental): Participants will receive 3 treatments of ELAPR002f injectable gel into the cheek area on each side of the face.
  Interventions: Device: ELAPR002f Injectable Gel
- Saline Active Control (Other): Participants will receive 3 treatments of Saline Active Control into the cheek area on each side of the face.
  Interventions: Other: Saline Active Control

INTERVENTIONS:
Device: ELAPR002f Injectable Gel — Intradermal Injections
  Arms: ELAPR002f Injectable Gel
Other: Saline Active Control — Intradermal Injections
  Arms: Saline Active Control

SUMMARY:
Visit the study website https://dawnacnescarstudy.com/ACT for more information. Atrophic acne scars are flat, indented or with an inverted center scars that develop at the endpoint of the normal healing process for acne. Acne scarring that remains after acne resolves has a significant impact on health related quality of life, including reduced self-esteem and embarrassment/self consciousness. ELAPR002f provides an immediate space-occupying effect for filling in the scar tissue. The purpose of this study is to assess how safe and effective ELAPR002f injectable gel is on adult participants with atrophic acne scars.

ELAPR002f Injectable Gel is an investigational device being developed for the treatment of facial atrophic acne scars. Participants are placed in 1 of 2 groups, called treatment arms. Each group receives a different treatment. There is a 1 in 4 chance that participants will be assigned to the saline active control group. Around 156 adult participants with moderate to severe atrophic acne scarring on both cheeks will be enrolled in the study in approximately 12 sites in Germany and Canada.

Participants will receive 3 treatments over 2 months of intradermal injections of either ELAPR002f injectable gel or saline active control and will be followed for up to an additional 12 months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participants in general good health, with no active COVID-19 infection, and seeking improvement of atrophic acne scars.
* Moderate to severe atrophic acne scarring (Grade 4 or 5 on the Allergan ASIS) on each cheek based on Evaluating Investigator's live assessment (both cheeks must qualify but do not need to have the same score) at the first screening visit.
* At least 5 rolling or boxcar-type acne scars in total within the predefined assessment field of either cheek in areas of otherwise normal healthy skin, as assessed by the treating investigator.

Exclusion Criteria:

* The participant has clinically significant acne on the face.
* Current cutaneous or mucosal inflammatory or infectious processes other than acne (eg, herpes), rosacea, abscess, an unhealed wound, or a cancerous or precancerous lesion, on the face.
* The participant presents with predominantly ice pick scars.
* History of keloid scar formation, hypertrophic scarring and/or post inflammatory hyperpigmentation or hypopigmentation.
* History of granulomatous or connective tissue disease.
* Diagnosed autoimmune disease (eg, Type 1 diabetes, rheumatoid arthritis, scleroderma, vitiligo).
* Diagnosed history of lung disease.
* Known hypersensitivity to the constituents of the device.
* Visual acuity of 20/100 or worse or abnormal confrontational visual fields or ocular motility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline in Acne Scar Area | Baseline to Day 181
  The acne scar area is calculated from 3D camera imaging software. Area is defined as the sum of the individual scar area of the 5 most prominent scars identified by the treating investigator (TI).
Number of Participants with Adverse Events | Up to Day 420
  An AE is defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory finding) in study participants, users, or other persons, whether or not related to the investigational medical device. This definition includes events related to the investigational medical device or comparator and events related to the procedures involved.
Number of Participants with Presence of Binding Antibodies | Up to Day 420
  Presence of binding antibodies
Number of Participants with Injection Site Responses (ISRs) and Systemic Responses | Up to Day 420
  Incidence of ISRs/systemic responses as recorded by e-diary for up to 30 consecutive days after each of the 3 treatment sessions starting on the day of injection. ISRs are defined as redness, pain after injection, tenderness to touch, firmness, swelling, lumps/bumps, bruising, itching and discoloration (not redness or bruising).
Number of Participants With Clinically Significant Changes From Baseline in Vital Sign Parameters | Up to Day 420
  Vital sign parameters include body temperature, systolic and diastolic blood pressure, pulse rate, and respiratory rate. The investigator will assess the results for clinical significance.
Number of Participants With Clinically Significant Changes From Baseline in Clinical Laboratory Parameters | Up to Day 420
  Clinical laboratory parameters include tests of hematology, chemistry, urinalysis and prolactin. The investigator will assess the results for clinical significance.
Number of Participants With Clinically Significant Changes From Baseline in Physical Measurements | Up to Day 420
  Physical measurements include weight and BMI. The investigator will assess the results for clinical significance.
Change from Baseline Procedure Pain | Up to Day 61
  Participants will assess procedure pain on an 11-point scale ranging from 0 (no pain) to 10 (worst pain imaginable) after each of the 3 treatment sessions.
Number of Participants with a Positive Skin Test | Up to Day 30
  Participants will undergo a skin test in the volar area of the forearm to test for hypersensitivity.
Number of Participants with Visual Disturbance Symptoms Associated with Vascular Occlusion | Up to Day 420
  Number of participants with any acute cognitive changes or any change in confrontational visual fields, ocular motility, or a worsening (1-line change or more) on the Snellen visual acuity assessment,

SECONDARY OUTCOMES:
Change from Baseline on the Overall Score of ACNE-Q Acne Scars Questionnaire | Up to Day 420
  The ACNE-Q Acne Scars questionnaire includes 10 questions that ask how much the participant is bothered by their acne scars on a 4-point scale ranging from 1=Not at all to 4=Very Much.
Change from Baseline on the Overall Score of ACNE-Q - Appearance-Related Distress | Up to Day 420
  ACNE-Q - Appearance-Related Distress questionnaire includes 8 questions that ask about how the participants describe themselves on a 4-point scale ranging from 1=Never to 4=Always.
Change from Baseline on the Overall Score of FACE-Q Satisfaction with Skin | Up to Day 420
  FACE-Q Satisfaction With Skin questionnaire includes 12 questions that ask how much the participants are satisfied or dissatisfied with their facial skin on a 4-point scale ranging from 1=Very Dissatisfied to 4=Very Satisfied.
Percentage of Participants Achieving "Responder" Status on Either Cheek Based on the Allergan Acne Scar Improvement Scale (ASIS), as assessed by the Evaluating Investigator | Up to Day 420
  A "responder" is a participant who achieves at least 1-grade improvement on either cheek based on the ASIS, as assessed by the EI. The ASIS is a 5-grade scale used to assess acne scar improvement ranging from 1=Almost None to 5=Severe. Each side of the face is scored separately.
Percentage of Participants who Achieve at Least a 20% Reduction in Acne Scar Area | Up to Day 420
  The acne scar area is calculated from 3D camera imaging software. Area is defined as the sum of the individual scar area of the 5 most prominent scars identified by the TI.
Percent Change from Baseline in Acne Scar Area | Up to Day 420
  The acne scar area is measured by 3D camera imaging software. Area is defined as the sum of the individual scar area of the 5 most prominent scars identified by the TI.
Percent Change from Baseline in Acne Scar Volume | Up to Day 420
  The acne scar volume is measured by 3D camera imaging software. Volume is defined as the sum of the individual scar volume of the 5 most prominent scars identified by the TI.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (12):
- Canada (7):
  - Alberta DermaSurgery Centre /ID# 243168, Edmonton, Alberta
  - Humphrey & Beleznay Cosmetic Dermatology /ID# 266634, Vancouver, British Columbia
  - Pacific Derm /ID# 227467, Vancouver, British Columbia
  - Dermetics Cosmetic Dermatology /ID# 227469, Burlington, Ontario
  - The Centre For Clinical Trials /ID# 233841, Oakville, Ontario
  - The Center For Dermatology /ID# 227470, Richmond Hill, Ontario
  - Bertucci MedSpa Inc. /ID# 227468, Woodbridge, Ontario
- Germany (5):
  - Hautok and Hautok-cosmetics /ID# 227474, Munich, Bavaria
  - Dermatologische Gemeinschaftspraxis Mahlow /ID# 262566, Blankenfelde-Mahlow, Brandenburg
  - Rosenpark Research /ID# 227471, Darmstadt, Hesse
  - MediCorium Zentrum fuer Dermatologie und Aesthetik /ID# 227475, Oberursel, Hesse
  - Privatpraxis Dr. Hilton & Partner /ID# 227472, Düsseldorf, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=2015-702-008